CLINICAL TRIAL: NCT00860704
Title: Intraoperative Goal Directed Fluid Therapy in Lean and Obese Patients
Brief Title: Goal Directed Fluid Therapy
Acronym: FLO1
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Andrea Holzer, MD, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EK 299/2006
Record Dates: First submitted 2009-03-11; First posted 2009-03-12 (Estimated); Last update posted 2018-10-18 (Actual); Status verified 2018-10

CONDITIONS: Goal Directed Fluid Therapy
Keywords: goal directed fluid therapy; lean patients; obese patients; crystalloids; Esophageal Doppler; tissue oxygenation; Fluid management during surgery; Fluid management
MeSH Terms: interventions — Ringer's Lactate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Ringerlactate lean (Active Comparator): fluidtherapy with crystalloids in lean patients
  Interventions: Drug: fluidotherapy with ringer-lactate
- Ringerlactate overweight (Active Comparator): fluidtherapy with crystalloids in overweight patients
  Interventions: Drug: fluidotherapy with ringer-lactate
- Ringerlactate obese (Active Comparator): fluidtherapy with crystalloids in obese patients
  Interventions: Drug: fluidotherapy with ringer-lactate

INTERVENTIONS:
Drug: fluidotherapy with ringer-lactate — a bolus of 250ml ringer-lactate is administered, if there is fluid demand monitored by the Esophageal Doppler

SUMMARY:
Intraoperative fluid demand will be monitored by Esophageal Doppler in lean and obese patients.

DETAILED DESCRIPTION:
To our knowledge no data are available on the effect of goal-directed fluid therapy on hemodynamics in lean patients and obese patients, respectively. Consequently, we want to compare lean patients (BMI <25) vs. obese patients (BMI >25) in regard of their respective needs for intraoperative fluid therapy, and the impact of the goal-directed fluid regimen on tissue oxygenation.

ELIGIBILITY:
Inclusion Criteria:

* female patients (18 - 80 years) undergoing elective gynecological open surgery (hysterectomy, ovarian cysts and tumors, myomectomy, endometriosis)

Exclusion Criteria:

* cardiac insufficiency (EF< 35%)
* renal insufficiency (creatinin clearance <30ml/min, dialysis)
* insulin dependant diabetes mellitus
* coagulopathy
* NYHA IV
* infection
* sepsis
* history of suspect malignant hyperthermia
* porphyria

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2007-11; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
different hemodynamic fluid responses in the different groups | every 10 minutes during surgery

SECONDARY OUTCOMES:
Subcutaneous oxygen tension (PsqO2) | every 10 minutes during surgery and 2 hours postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Holzer, MD, Principal Investigator — Medical University Vienna, Department of Anesthesiology and General Intensive Care Medicine
Locations (1):
- Medical University Vienna, Vienna, Austria

REFERENCES:
- [Background] Gan TJ, Soppitt A, Maroof M, el-Moalem H, Robertson KM, Moretti E, Dwane P, Glass PS. Goal-directed intraoperative fluid administration reduces length of hospital stay after major surgery. Anesthesiology. 2002 Oct;97(4):820-6. doi: 10.1097/00000542-200210000-00012. PMID 12357146